CLINICAL TRIAL: NCT05604716
Title: An Observational Cross-sectional Follow-up Study on Digestive Physiological and Social Philosophical Functions of Solid Pseudopapillary Neoplasm of the Pancreas (SPN)
Brief Title: Cross-sectional Follow-up on Digestive and Social Functions of SPN
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Qiaofei Liu, clinical chief professor, Peking Union Medical College Hospital
Other Study IDs: S-K1034
Record Dates: First submitted 2022-10-10; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Solid Pseudopapillary Tumor of the Pancreas; Pancreas Cancer
Keywords: Solid Pseudopapillary Neoplasm of the Pancreas; surgery; follow up; digestive physiological function; social psychological function
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SPN patients
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
An observational cross-sectional follow-up study on the quality of life (two aspects, digestive physiological and social psychological functions) of solid pseudopapillary neoplasm of the pancreas (SPN) patients recruited in PUMCH from 2001 to 2026. The quality of life is evaluated by a questionnaire made up of eight validated scales.

DETAILED DESCRIPTION:
Solid pseudopapillary neoplasm of the pancreas (SPN) is a rare tumor with uncertain malignant potential. It is a rare entity of pancreatic tumor with low potential malignancy, constituting 1% to 3% of pancreatic tumors and 10%-15% of pancreatic cystic neoplasm. Although the reported cases of SPN have been increasing rapidly all over the world during the last two decades, its long-term follow-up studies in large cohorts remain missing.

From this, this observational cross-sectional follow-up study on the digestive physiological and social psychological functions of SPN patients aims to achieve a comprehensive understanding on how SPN and surgery affects the quality of life. Patients are recruited in PUMCH from 2001-2026 with a definite pathological diagnosis.

The quality of life after surgery is evaluated by a questionnaire made up of six validated scales (digestive physiological functions via: 8 symptoms scale of the EORTC core quality of life questionnaire (EORTC QLQ-C30); gastrointestinal symptom rating scale questionnaire (GSRS); social psychological functions via: sense of coherence-9 questionnaire (SOC-9); patient health questionnaire-9 questionnaire (PHQ-9), general anxiety disorder-7 questionnaire (GAD-7) ; post-traumatic embitterment disorder 21 questionnaire (PTED-21); work ability index questionnaire (WAI); body image scale questionnaire (BIS)). To our knowledge, this is the largest SPN cohort worldwide and the first study to concentrate on the quality of life of SPN after operations.

ELIGIBILITY:
Inclusion Criteria:

* SPN patients with pathological diagnosis after surgery
* Approval to participate
* patients with valid and complete questionnaires results inspected by two experienced surgeons

Exclusion Criteria:

* Refusal to participate
* patients with invalid or incomplete questionnaires results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All of the hospitalized patients of SPN with a definite pathological diagnosis who underwent operations from 2001 to 2026 in Peking Union Medical College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2001-01-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
scores of digestive physiological and social psychological functions | up to 15 years after surgery
  The primary outcome is a score of digestive physiological and social psychological functions of SPN patients up to 15 years after surgery. The score is evaluated by a follow-up questionnaire made up of: digestive physiological functions via 8 symptoms scale of the EORTC core quality of life questionnaire and gastrointestinal symptom rating scale questionnaire; social psychological functions via sense of coherence-9, patient health questionnaire-9, general anxiety disorder-7; post-traumatic embitterment disorder 21; work ability index questionnaire, body image scale.R aw scores will undergo a linear transformation for standardization. The maximum and minimum score is 100 and 0, respectively. Higher scores on the digestive physiological and social psychological functioning scales represent better quality of life, whereas higher scores on the symptom scale represent more serious symptoms or poorer quality of life.

SECONDARY OUTCOMES:
progressive-free survival | the time from the surgery to the progressive conditions (From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to up 180 months)
  the time from the surgery to the progressive conditions (from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to up 180 months)

CONTACTS AND LOCATIONS:
Overall Officials: Qiaofei Liu, Study Chair — Department of General Surgery, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No